CLINICAL TRIAL: NCT01448863
Title: Metabolomic Embryo Profiles of Obese in Vitro Fertilization (IVF) Patients and Their Relationship With Polycystic Ovary Syndrome (PCO)
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Jose Bellver, Gynecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: 1005-C-070-JB
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Infertility; Obesity
MeSH Terms: conditions — Infertility; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- CONTROL: Fertile women (egg-donors)
  Interventions: Other: Culture medium metabolomic analysis
- WITH PCO: Obese women with Polycystic Ovarian Syndrome
  Interventions: Other: Culture medium metabolomic analysis
- NO PCO: Obese women without Polycystic Ovarian Syndrome
  Interventions: Other: Culture medium metabolomic analysis

INTERVENTIONS:
Other: Culture medium metabolomic analysis — During the embryo transfer at day 3, the investigators keep and freeze a small drop of the culture medium of each embryo transferred. Each drop of culture medium will have a volume of 40-50 microliters, before freezing is spun at 10.000 rps to avoid any possible contamination.
  The frozen media culture is analyzed for the metabolomic profile.

SUMMARY:
The present study aims to elucidate if there is a metabolomic profile alteration in the embryos of obese women in order to understand if the reduced implantation rate observed in these patients is directly related to this factor. Furthermore, the investigators seek to establish if there is any difference between obese women with Polycystic Ovary Syndrome (PCO) and without PCO. The investigators compare these metabolomic profile embryos with embryos of egg-donation programme.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30 kg/m2
* Age < 38 years old
* Non smokers
* First IVF cycle (groups 2 & 3, not Control group)
* Normal uterus (seen by ultrasound)
* normal basal hormonal profile(FSH,LH,estradiol,testosterone,androstenedione, insulin, SHBG, glucose, AMH)
* Antral follicle count(> 5 FA for each ovary)
* Menses every 25-35 days.

Exclusion Criteria:

* < 5 or > 20 oocytes retrieved after stimulation cycle
* estradiol >3000 pg/ml or progesterone > 1,5 ng/ml on the hCG day.
* < 2 evolutive embryos in the culture medium.

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 45 women divided into three groups: A)15 Obese women without Polycystic Ovarian Syndrome: BMI > 30 kg/m2 , age < 38 years old, normal basal hormonal profile (FSH, LH, estradiol, testosterone, androstenedione, insulin, SHBG, glucose, AMH, and antral follicle count(> 5 FA for each ovary), menses every 25-35 days.
  B)15 Obese women with Polycystic Ovarian Syndrome: BMI > 30 kg/m2, age < 38 years old, basal hormonal profile with or without hyperandrogenism and ultrasound ovary aspect of PCO.
  C)15 Fertile women (egg-donors): BMI 20-24.9 kg/m2. All the patients have normal uterine conditions, are not smokers, without endometriosis or hidrosalpinx. All the male partners have sperm parameters: count(> 5 mill/ml,15% motility,> 0% normal morphology)and BMI < 28 kg/m2.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Metabolic profile of culture media of Day 3 embryos | 3 days
  Determine differences in the metabolomic profile of the culture media of day 3 embryos, obtained after in vitro fertilization, according to the presence of obesity associated or not with polycystic ovary syndrome.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - IVI Valencia, Valencia, Valencia
  - IVI Valencia, Valencia

REFERENCES:
- [Derived] Bellver J, De Los Santos MJ, Alama P, Castello D, Privitera L, Galliano D, Labarta E, Vidal C, Pellicer A, Dominguez F. Day-3 embryo metabolomics in the spent culture media is altered in obese women undergoing in vitro fertilization. Fertil Steril. 2015 Jun;103(6):1407-15.e1. doi: 10.1016/j.fertnstert.2015.03.015. Epub 2015 Apr 29. PMID 25935493